CLINICAL TRIAL: NCT06211595
Title: To Evaluate the Safety and Feasibility of the DragonFire Transcatheter Radiofrequency Myocardial Ablation System
Brief Title: Feasibility Study of the DragonFire for Hypertrophic Obstructive Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hangzhou Valgen Medtech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DragonFire-01
Record Dates: First submitted 2024-01-09; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The treament of DragonFire Transcatheter myocardial ablation system (Experimental): If drug therapy does not work or drug side effects are not tolerated, transaortic interventional surgery can be evaluated
  Interventions: Device: DragonFire Transcatheter Myocardial Radiofrequency Ablation System

INTERVENTIONS:
Device: DragonFire Transcatheter Myocardial Radiofrequency Ablation System — The patients with hypertrophic obstructive cardiomyopathy were treated with a transcatheter myocardial radiofrequency ablation system and its guiding system under the guidance of echocardiography

SUMMARY:
This is a prospective, single-center, single-arm clinical study. All patients were diagnosed with obstructive hypertrophic cardiomyopathy, and only subjects who met the instrument indications of this study were treated. After signing an informed consent form, subjects are enrolled and treated with the DragonFire Transcatheter Myocardial Ablation System. All subjects receive clinical follow-up immediately after the procedure, before discharge, 30 days after the procedure, 6 months after the procedure, and 12 months after the procedure.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm clinical study. All patients were diagnosed with obstructive hypertrophic cardiomyopathy, and only subjects who met the instrument indications of this study were treated. After signing an informed consent form, subjects are enrolled and treated with the DragonFire Transcatheter Myocardial Ablation System. The primary efficacy endpoint was the rate of major adverse events 30 days after surgery. The safety endpoints were the rate of immediate postoperative success and postoperative device success All subjects receive clinical follow-up immediately after the procedure, before discharge, 30 days after the procedure, 6 months after the procedure, and 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Obstructive hypertrophic cardiomyopathy, peak LVOT pressure difference ≥50mmHg at rest or after excitation;
3. Obvious clinical symptoms, fatigue, shortness of breath, fatigue angina pectoris, syncope, etc., seriously affect the quality of life, and adequate drug treatment is not effective or can not tolerate drug side effects, after evaluation, transaortic interventional surgery can be performed;

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant;
2. interventricular septum thickness ≥30mm;
3. non-hypertrophic obstructive cardiomyopathy;
4. Presence of cardiac neoplasms;
5. A history of interventricular septal resection or alcohol ablation, or Liwen surgery;
6. Combined with other heart diseases requiring surgical treatment;
7. Heart failure (after intensive anti-heart failure treatment, there are still symptoms of resting heart failure, such as left ventricular ejection fraction < 50%, N-terminal -B type natriuretic peptide precursor, NT-pro BNP≥5000pg/ml, pulmonary edema, pleura or pericardial effusion, etc.);
8. Significant coronary lesions, or borderline lesions, requiring coronary revascularization due to mismatch between coronary perfusion and demand (QFR or FFR < 0.8), or coronary ischemic events within 30 days;
9. Bleeding diseases or clotting disorders; Or there is a contraindication of antithrombotic drug therapy;
10. estimated Glomerular Filtration Rate (eGFR) < 35ml/min;
11. Life expectancy was less than 12 months, and the investigator judged that the patient had poor compliance and could not complete the study as required; Or other circumstances in which the investigator considers the subject unsuitable for the study;
12. Subject is currently participating in an investigational drug or device study that has not completed its primary endpoint or that would clinically interfere with the endpoint of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of MAE | 30 days
  Major adverse Event (MAE) is defined as any instrument-related or surgery-related complication, including death, emergency surgery, severe pericardial tamponade requiring pericardiocentesis or surgery, bleeding, surgery-related stroke, pacemaker implantation, and mechanically assisted circulation

SECONDARY OUTCOMES:
Acute procedural success | Immediately after procedure
  The device arrived at the intended treatment site for ablation, and was successfully withdrawn after ablation
Percentage of subjects with left ventricular outflow tract pressure (LVOTG) reduction of ≥50% or left ventricular outflow tract pressure (LVOTG) < 30mmHg | 12 months
  Percentage of subjects with left ventricular outflow tract pressure (LVOTG) reduction of ≥50% or LVOTG< 30mmHg after the procedure
Incidence of device or device-related adverse events and device defects | 12 months
Quality of life improvement | 6 months, 12months
  Improvement in quality of life (QoL) , as measured by the Kansas City Cardiomyopathy Questionnaire，a scale of 0-100 with higher scores indicating better health

CONTACTS AND LOCATIONS:
Overall Officials: Fang ZhenFei, Phd, Principal Investigator — The Second Xiangya Hospital, Central South University
Locations (1):
- The Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No